CLINICAL TRIAL: NCT05569733
Title: Simultaneous Fluorodeoxyglucose and Magnetic Resonance Imaging (18F-FDG PET/MR) Study of Metabolic and Structural Changes in Visual Snow Syndrome Compared to Healthy Controls
Brief Title: Simultaneous Fluorodeoxyglucose Positron Emission Tomography (PET) and Magnetic Resonance (MR) in Visual Snow Syndrome
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S58764-S58571
Record Dates: First submitted 2022-09-27; First posted 2022-10-06 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2022-09

CONDITIONS: Visual Snow Syndrome
Keywords: FDG PET; PET/MR; volumetry; visual analysis; discriminant analysis
MeSH Terms: conditions — visual snow syndrome | interventions — Positron-Emission Tomography; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VSS: Patients with visual snow syndrome
  Interventions: Diagnostic Test: simultaneous fluor-18 fluorodeoxyglucose (FDG) positron emission tomography with magnetic resonance imaging (PET/MRI)
- controls: healthy, screened age-matched controls
  Interventions: Diagnostic Test: simultaneous fluor-18 fluorodeoxyglucose (FDG) positron emission tomography with magnetic resonance imaging (PET/MRI)

INTERVENTIONS:
Diagnostic Test: simultaneous fluor-18 fluorodeoxyglucose (FDG) positron emission tomography with magnetic resonance imaging (PET/MRI) — All subjects fast at least for 4 hours prior to 18F-FDG injection. 18F-FDG is injected intravenously (150 megabecquerel (MBq)) in standard ambient conditions, supine in a dark, noise free room with eyes and ears open. 18F-FDG PET images are acquired for 20 min on a simultaneous GE Signa 3 Tesla (3T) PET/MR scanner with integrated Time-of-Flight (TOF) (GE Healthcare, Chicago, USA). Simultaneous with the 18F-FDG PET/MR acquisition, zero-echo-time (ZTE) MR data are acquired for attenuation correction and a 3D volumetric T1-weighted BRAVO MR sequence using a vendor supplied high-resolution 8-channel phased array head coil (GE Healthcare, Milwaukee, USA).

SUMMARY:
Visual snow syndrome (VSS) is a neurologic condition where patients experience tiny flickering dots in their entire visual field. It has been reported that the brain consumes more glucose in the lingual gyrus (a subdivision of the occipital cortex) and that this also shows increased volume of grey matter (neurons and supporting cells). In this study, the investigators apply fluor-18 fluorodeoxyglucose positron emission tomography with magnetic resonance imaging (18F-FDG PET/MR) in patients with VSS and compare this to healthy controls. Aside from an analysis in each brain volume element (voxel), the accuracy of classifying groups based on a volume-of-interest (VOI) analysis of both PET and MR is studied, Lastly, this is also compared to a visual assessment of the PET and MR images.

DETAILED DESCRIPTION:
Aim : Prospective measurement of brain glucose metabolism and structural integrity in the brain of subjects with visual snow syndrome (VSS). Voxel-based and volume-of interest comparison to age matched healthy controls retrospectively obtained on the same simultaneous PET/MR imaging system.

Hypothesis : 1/ VSS patients show overactivation of parts of the visual system, in particular the lingual gyrus, which is likely related to larger volume of the gyrus on structural imaging. 2/ Discrimination of VSS patients versus controls can be done by visual read of FDG PET and/or volume-of-interest based discriminant analysis.

Methods : Recruitment through neurology practice specialised in VSS, detailed history taking and assessment of in/exclusion criteria, scanning with simultaneous18F-FDG PET/MR Signa GE Healthcare.

Analysis : visual assessment, group-based voxel and volume-of-interest based analysis (FDG PET, volumetry T1 MRI) with appropriate statistics and corrections for multiple regional comparisons. Discriminant analysis on VOI based data. Dual observer scoring of visual data and assessment of accuracy, sensitivity and specificity of visual image analysis compared to clinical final diagnosis.

ELIGIBILITY:
GROUP 1: VSS Patients

Inclusion Criteria:

* M/F, age 18-85,
* diagnosis of VSS by an experienced neurologist : dynamic, continuous, black and white tiny dots in the entire visual field lasting longer than 3 months, with at least two additional visual symptoms

Exclusion Criteria:

- other underlying neurological conditions inclusive ophthalmological examinations

GROUP 2 : Controls

Inclusion Criteria:

* age 18-85 years, M/F, in general healthy condition
* normal neurological examination, Mini-Mental State Examination (MMSE) ≥ 28, Beck's Depression Inventory (BDI) score ≤ 9, and a normal structural volumetric MRI.

Exclusion Criteria:

* history of major internal pathology, neurological and/or psychiatric disorders (including psychosis, depression, and anxiety),
* history of frequent migraine attacks, substance abuse or current use of any central acting medication
* first-degree relatives with dementia.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1 : Visual Snow Syndrome patients Group 2 : Healthy Controls
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2017-09-02 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Group difference in regional brain metabolism as assessed with 18F-FDG positron emission tomography | analysis done immediately after imaging
  Visual, voxel- and volume-of-interest based assessment of of FDG PET
Group difference in regional brain volume assessed with volumetric magnetic resonance imaging. | at baseline
  Visual, voxel- and volume-of-interest based assessment of MRI images

SECONDARY OUTCOMES:
Discriminant analysis of PET metabolic differences | at baseline
  Statistical discriminant analysis of FDG between VSS patients and controls
Visual scoring of PET metabolic differences | at baseline
  Visual scoring of FDG between VSS patients and controls
Discriminant analysis of MR volumetric differences | at baseline
  Statistical discriminant analysis of regional MR volumetry between VSS patients and controls
Visual scoring of MR volumetric differences | at baseline
  Visual scoring of regional MR volumetry between VSS patients and controls

CONTACTS AND LOCATIONS:
Overall Officials: Koen Van Laere, MD PhD, Principal Investigator — Head Nuclear Medicine, University Hospitals Leuven

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared on a reasonable request, including full FDG PET and MRI data as well as supporting information.
Supporting Information: Study Protocol, ICF
Access Criteria: Contact PI by email.

REFERENCES:
- [Derived] Van Laere K, Ceccarini J, Gebruers J, Goffin K, Boon E. Simultaneous 18F-FDG PET/MR metabolic and structural changes in visual snow syndrome and diagnostic use. EJNMMI Res. 2022 Dec 30;12(1):77. doi: 10.1186/s13550-022-00949-0. PMID 36583806